CLINICAL TRIAL: NCT00946894
Title: Five-year Follow up of a Randomized Clinical Trial of Total Thyroidectomy Versus Dunhill Operation Versus Bilateral Subtotal Thyroidectomy for Multinodular Non-toxic Goiter.
Brief Title: Outcomes of Different Thyroid Resections for Multinodular Non-toxic Goiter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Piotr Laider / Head of the Biomedical Research Committee of the Jagiellonian University, Jagiellonian University Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBN/501/ZKL/68/L
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Goiter
Keywords: Total thyroidectomy; Subtotal thyroidectomy; Dunhill operation; Recurrent nodular goiter; Completion thyroidectomy; Recurrent laryngeal nerve palsy; Hypoparathyroidism following thyroidectomy; Recurrent goiter
MeSH Terms: conditions — Goiter; Goiter, Nodular; Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Total thyroidectomy (Experimental): Patients who underwent total thyroidectomy
  Interventions: Procedure: Total thyroidectomy
- Dunhill operation (Experimental): Patients who underwent unilateral total thyroid lobectomy and contralateral subtotal thyroid lobectomy
  Interventions: Procedure: Dunhill operation
- Bilateral subtotal thyroidectomy (Active Comparator): Patients who underwent bilateral subtotal thyroidectomy
  Interventions: Procedure: Bilateral subtotal thyroidectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — Total thyroidectomy
  Other Names: TT
  Arms: Total thyroidectomy
Procedure: Dunhill operation — Unilateral total thyroid lobectomy and contralateral subtotal thyroid lobectomy
  Other Names: DO
  Arms: Dunhill operation
Procedure: Bilateral subtotal thyroidectomy — Bilateral subtotal thyroidectomy
  Other Names: BST
  Arms: Bilateral subtotal thyroidectomy

SUMMARY:
The aim of this three-arm randomized study was to evaluate results of different thyroid resection modes among patients with bilateral multinodular non-toxic goiter, with special emphasis put on recurrence rate and morbidity rate, in a 5-year follow-up.

DETAILED DESCRIPTION:
The extent of thyroid resection in bilateral multinodular non-toxic goiter remains controversial. Surgeons still continue to debate whether the potential benefits of total thyroidectomy outweigh the potential complications. Most low-volume surgeons avoid to perform total thyroidectomy owing to the possible complications such as permanent recurrent laryngeal nerve palsy and permanent hypoparathyroidism. On the other hand, the increasing number of total thyroidectomies are currently performed in high-volume endocrine surgery units, and the indication for this procedure include thyroid cancer, Graves disease and multinodular goiter. Recently there has been increasing acceptance for performing total thyroidectomy for bilateral multinodular non-toxic goiter as it removes the disease process completely, lowers local recurrence rate and avoids the substantial risk of reoperative surgery, and involves only a minimal risk of morbidity. This common perception is based largely on single-institution retrospective data, a few multi-institutional retrospective experiences, and only a few prospective randomized studies comparing the outcomes of total vs. subtotal thyroidectomy.

ELIGIBILITY:
Inclusion Criterion

* a bilateral non-toxic multinodular goiter with normal appearing on ultrasound of the neck posterior aspects of both thyroid lobes.

Exclusion Criteria:

* multinodular goiter involving posterior aspect/s of thyroid lobe/s,
* suspicion of thyroid cancer,
* previous thyroid surgery,
* thyroiditis,
* subclinical or clinically overt hypothyroidism or hyperthyroidism,
* pregnancy or lactation,
* age < 18 years or > 65 years,
* ASA 4 grade (American Society of Anesthesiology),
* inability to comply with the follow-up protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2000-01; Primary Completion 2003-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was prevalence of recurrent goiter and need for redo surgery. | at 12, 24, 36, 48 and 60 months after surgery

SECONDARY OUTCOMES:
Secondary outcome measure was postoperative morbidity rate (hypoparathyroidism and recurrent laryngeal nerve injury). | at 3, 6, 9, 12, 24, 36, 48 and 60 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University College of Medicine
Locations (1):
- Jagiellonian University, College of Medicine, Department of Endocrine Surgery, 3rd Chair of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Snook KL, Stalberg PL, Sidhu SB, Sywak MS, Edhouse P, Delbridge L. Recurrence after total thyroidectomy for benign multinodular goiter. World J Surg. 2007 Mar;31(3):593-8; discussion 599-600. doi: 10.1007/s00268-006-0135-0. PMID 17308855
- [Background] Wheeler MH. Total thyroidectomy for benign thyroid disease. Lancet. 1998 May 23;351(9115):1526-7. doi: 10.1016/S0140-6736(05)61116-6. No abstract available. PMID 10326531
- [Background] Ozbas S, Kocak S, Aydintug S, Cakmak A, Demirkiran MA, Wishart GC. Comparison of the complications of subtotal, near total and total thyroidectomy in the surgical management of multinodular goitre. Endocr J. 2005 Apr;52(2):199-205. doi: 10.1507/endocrj.52.199. PMID 15863948
- [Background] Moalem J, Suh I, Duh QY. Treatment and prevention of recurrence of multinodular goiter: an evidence-based review of the literature. World J Surg. 2008 Jul;32(7):1301-12. doi: 10.1007/s00268-008-9477-0. PMID 18305998
- [Background] Tezelman S, Borucu I, Senyurek Giles Y, Tunca F, Terzioglu T. The change in surgical practice from subtotal to near-total or total thyroidectomy in the treatment of patients with benign multinodular goiter. World J Surg. 2009 Mar;33(3):400-5. doi: 10.1007/s00268-008-9808-1. PMID 18958517
- [Background] Agarwal G, Aggarwal V. Is total thyroidectomy the surgical procedure of choice for benign multinodular goiter? An evidence-based review. World J Surg. 2008 Jul;32(7):1313-24. doi: 10.1007/s00268-008-9579-8. PMID 18449595
- [Background] Phitayakorn R, McHenry CR. Follow-up after surgery for benign nodular thyroid disease: evidence-based approach. World J Surg. 2008 Jul;32(7):1374-84. doi: 10.1007/s00268-008-9487-y. PMID 18311576
- [Background] Barczynski M, Konturek A, Cichon S. Randomized clinical trial of visualization versus neuromonitoring of recurrent laryngeal nerves during thyroidectomy. Br J Surg. 2009 Mar;96(3):240-6. doi: 10.1002/bjs.6417. PMID 19177420
- [Derived] Barczynski M, Konturek A, Hubalewska-Dydejczyk A, Golkowski F, Nowak W. Ten-Year Follow-Up of a Randomized Clinical Trial of Total Thyroidectomy Versus Dunhill Operation Versus Bilateral Subtotal Thyroidectomy for Multinodular Non-toxic Goiter. World J Surg. 2018 Feb;42(2):384-392. doi: 10.1007/s00268-017-4230-1. PMID 28942461
- [Derived] Barczynski M, Konturek A, Hubalewska-Dydejczyk A, Golkowski F, Cichon S, Nowak W. Five-year follow-up of a randomized clinical trial of total thyroidectomy versus Dunhill operation versus bilateral subtotal thyroidectomy for multinodular nontoxic goiter. World J Surg. 2010 Jun;34(6):1203-13. doi: 10.1007/s00268-010-0491-7. PMID 20174803